CLINICAL TRIAL: NCT03032965
Title: Adenosine Study in Paroxysmal Atrial Fibrillation
Brief Title: Adenosine to Assess Complete Conduction Block During Catheter Ablation of Paroxysmal Atrial Fibrillation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Hamid Ghanbari, Assistant Professor of Internal Medicine, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HUM00048922
Record Dates: First submitted 2016-09-01; First posted 2017-01-26 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2017-12-13 (Actual); Status verified 2017-11

CONDITIONS: Atrial Fibrillation
Keywords: atrial fibrillation; ablation; adenosine
MeSH Terms: conditions — Atrial Fibrillation | interventions — Adenosine; Isoproterenol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Adenosine and Isoproterenol (Experimental): Patients in this group will receive 12-24mg of adenosine for each PV in order to assess dormant PV conduction.
  Interventions: Drug: Adenosine; Drug: Isoproterenol
- Isoproterenol (Other): This group will not receive adenosine during the procedure.
  Interventions: Drug: Isoproterenol

INTERVENTIONS:
Drug: Adenosine — Subject will receive 6-24 mg of intravenous adenosine given rapidly for each PV in order to assess dormant PV conduction.
  Subjects in this group will also receive isoproterenol to assess inducibility of AF with re-isolation of PVs and targeting non PV sources of AF if necessary.Isoproterenol will be infused through a femoral vein at rates of 5, 10, 15, and 20 μg/min for 2 minutes at each infusion rate.
  Arms: Adenosine and Isoproterenol
Drug: Isoproterenol — Isoproterenol will be infused through a femoral vein at rates of 5, 10, 15, and 20 μg/min for 2 minutes at each infusion rate. The isoproterenol infusion will be discontinued upon induction of AF, a decrease in systolic blood pressure to<85 mmHg, complaints of severe chest tightness, electrocardiographic changes suggestive of ischemia, or upon completion of the infusion protocol.
  Other Names: Isuprel

SUMMARY:
The purpose of this study is to determine if additional ablation during the first procedure as the result of the ability to medically induce quiet atrial arrhythmias will improve clinical outcome in patients with atrial fibrillation thus decreasing the need for additional ablation procedures.

DETAILED DESCRIPTION:
Hypothesis:

1. Adenosine reveals incomplete conduction block due to partial tissue injury/stunning during catheter ablation of atrial fibrillation.
2. Identification of incomplete conduction block by adenosine improves clinical outcomes including an increase in efficacy and a decrease in need for repeat procedures after catheter ablation of atrial fibrillation.

Objectives:

1. In patients with paroxysmal Atrial Fibrillation (AF), the prevalence of Pulmonary Vein (PV) reconnection during adenosine infusion after complete PV isolation using conventional techniques will be determined.
2. Patients will be randomized to further ablation to achieve complete isolation during adenosine infusion vs to no further ablation.
3. Primary endpoint of the study will be freedom from any atrial arrhythmias 6 months after a single ablation procedure in the absence of antiarrhythmic drug therapy.
4. Secondary endpoints will include number of repeat ablation procedures because of documented recurrence of symptomatic AF or atrial flutter/tachycardia, outcome after 2 ablation procedures; Proportion of patients with AF or atrial flutter/tachycardia occuring during the first three months post ablation, prevalence of recovery of conduction into PVs during repeat ablation procedures in both groups, procedure duration, and incidence of peri-procedural complications including stroke, PV stenosis, cardiac perforation, atrio-esophageal fistulae, and death.

ELIGIBILITY:
Inclusion Criteria:

1. Patients >18 and <75 who are able to give informed consent undergoing atrial fibrillation ablation procedure.
2. Paroxysmal Atrial fibrillation lasting = 7 days which is self-terminating. It is considered recurrent if two or more episodes occur.
3. Failure or unwilling to take class I or III anti-arrhythmic drugs

Exclusion Criteria:

1. History of asthma
2. Patients with severe coronary artery disease, stable/unstable angina, or ongoing myocardial ischemia
3. Previous cardiac surgery ( excluding CABG and mitral valve surgery)
4. Symptomatic congestive heart failure including but not limited to NYHA III/IV and/or documented ejection fraction <40% measured by acceptable cardiac testing,
5. Left atrial diameter >55mm
6. Moderate to severe mitral or aortic valve disease
7. Myocardial infarction within three months of enrollment
8. Congenital heart disease where it increases the risk of an ablative procedure
9. Prior ASD/PFO closure with a device using a percutaneous approach
10. Hypertrophic cardiomyopathy (LV wall thickness >1.5mm)
11. Pulmonary Hypertension (mean or systolic PA pressure> 50mmHg on Doppler echocardiography
12. Any prior ablation of atrial fibrillation
13. Enrollment in any other arrhythmia protocol
14. Any ventricular arrhythmia being treated where the arrhythmia or management may interfere with this study
15. Active infection or sepsis
16. Any history of cerebrovascular disease including stroke or TIAs
17. Pregnancy or lactation
18. Left atrial thrombus at the time of ablation
19. Untreatable allergy to contrast media
20. Any diagnosis of atrial fibrillation secondary to electrolyte disturbance, thyroid disease, or any other reversible or non-cardiovascular causes
21. History of blood clotting(bleeding or thrombotic) abnormalities
22. Known sensitivities to heparin or warfarin
23. Severe COPD (defined as FEV1 <1)
24. Severe comorbidity or poor general physical/mental health that, in opinion of the investigator, will not allow the patient to be a good study candidate (i.e. other disease processes, mental capacity, substance abuse, shortened life expectancy)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 131 (Actual)
Dates: Start 2011-10; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hamid Ghanbari, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Two subjects were not randomized.
Groups:
- Adenosine and Isoproterenol: Patients in this group will receive 12-24mg of adenosine for each PV in order to assess dormant PV conduction.
  Adenosine: Subject will receive 6-24 mg of intravenous adenosine given rapidly for each PV in order to assess dormant PV conduction.
  Subjects in this group will also receive isoproterenol to assess inducibility of AF with re-isolation of PVs and targeting non PV sources of AF if necessary.Isoproterenol will be infused through a femoral vein at rates of 5, 10, 15, and 20 μg/min for 2 minutes at each infusion rate.
  Isoproterenol: Isoproterenol will be infused through a femoral vein at rates of 5, 10, 15, and 20 μg/min for 2 minutes at each infusion rate. The isoproterenol infusion will be discontinued upon induction of AF, a decrease in systolic blood pressure to<85 mmHg, complaints of severe chest tightness, electrocardiographic changes suggestive of ischemia, or upon completion of the infusion protocol.
Period: Overall Study
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Started | 61 | 68
Completed | 61 | 68
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adenosine and Isoproterenol | Isoproterenol | Total
Number analyzed (Participants) | 61 | 68 | 129
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.7 (8.7) | 58.9 (10.7) | 59.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24 | 15 | 39
  Male | 37 | 53 | 90
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 61 | 68 | 129
Left ventricular ejection fraction [Mean (Standard Deviation); unit: Percentage] | 59.7 (5.4) | 59.3 (5.6) | 59.5 (7.8)
left atrial diameter [Mean (Standard Deviation); unit: milli meters] | 41.0 (5.3) | 41.2 (6.4) | 41.1 (8.3)
Hypertension [Count of Participants; unit: Participants] — Participants with a documented history of hypertension or being treated for hypertension with medications
  Participants | 33 | 28 | 61
Diabetes Mellitus [Count of Participants; unit: Participants] — participants with a history of diabetes mellitus or current treatment for diabetes
  Participants | 6 | 8 | 14
Obstructive sleep apnea [Count of Participants; unit: Participants] — participants with a history of obstructive sleep apnea
  Participants | 15 | 19 | 34
Cerebrovascular accident [Count of Participants; unit: Participants] — participants with a history of cerebrovascular accident
  Participants | 2 | 4 | 6
Repeat procedure [Count of Participants; unit: Participants] — These are patients who had a previous ablation prior to entering the study
  Participants | 20 | 23 | 43
CHADS2 Score ( Congestive heart failure, Hypertension, Age > 75 years, Diabetes Mellitus, Stroke [Mean (Standard Deviation); unit: units on a scale] — Each of these five variables is given 1 point for its presence, except stroke is given 2 points. Each individual point is added, so the score ranges possible are 0 to 6 where 0 represents no risk factors and 6 represents highest number of risk factors.
  units on a scale | 0.8 (0.7) | 0.7 (0.7) | 0.75 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Any Atrial Arrhythmias
Description: Primary endpoint of the study will be number of participants who are free from any atrial arrhythmias after a single ablation procedure in the absence of antiarrhythmic drug therapy
Time Frame: 2- 14 months after Ablation procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 61 | 68
Participants | 24 | 23
Statistical Analysis 1: Comparison: Adenosine and Isoproterenol vs Isoproterenol; Test type: Superiority; p = .83, Log Rank; Kaplan Meier log rank

2. Secondary Outcome: Number of Subjects Who Need Repeat Ablations
Description: Number of participants who had one or more repeat ablation procedures due to documented recurrence of Symptomatic AF or atrial flutter/tachycardia.
Time Frame: date of ablation to 6 months after procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 61 | 68
Participants | 12 | 9
Statistical Analysis 1: Comparison: Adenosine and Isoproterenol vs Isoproterenol; Test type: Superiority; p = .35, t-test, 2 sided

3. Secondary Outcome: Number of Subjects With AF or Atrial Flutter/Tachycardia Occurring During the First Three Months Post Ablation
Time Frame: first three months post ablation
Population: This data was not collected.
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Pulmonary Veins That Recovered Conduction During Repeat Ablation Procedures in Both Groups
Description: Prevalence of recovery of conduction into pulmonary veins during repeat ablation procedures in both groups. This is determined by surgeon assessment using a circular mapping catheter to identify recovery of conduction into the pulmonary veins.
Time Frame: post-procedure (6 months)
Population: Only 21 participants had repeat ablations; each participant has four pulmonary veins therefore the number of connections measured is based 4 x the number of participants
Measure: Count of Units; unit: pulmonary veins
Units Other Than Participants: pulmonary veins
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 12 | 9
Number analyzed (pulmonary veins) | 48 | 36
pulmonary veins | 29 | 28
Statistical Analysis 1: Comparison: Adenosine and Isoproterenol vs Isoproterenol; Test type: Superiority; p = 0.09, t-test, 2 sided

5. Secondary Outcome: Incidence of Stroke
Description: Number of subjects who develop stroke within 30 days after procedure.
Time Frame: peri-procedural (0 to 30 days after procedure)
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 61 | 68
Participants | 0 | 0

6. Secondary Outcome: Incidence of Pulmonary Vein Stenosis
Description: Number of subjects who develop Symptomatic pulmonary vein stenosis
Time Frame: 6 months post-procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 61 | 68
Participants | 0 | 0

7. Secondary Outcome: Incidence of Cardiac Perforation
Description: Number of subjects who develop perforation of heart during ablation
Time Frame: within 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 61 | 68
Participants | 0 | 0

8. Secondary Outcome: Incidence of Atrio-esophageal Fistula
Description: Number of subjects who develop connection between heart and the esophagus
Time Frame: within 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 61 | 68
Participants | 0 | 0

9. Secondary Outcome: Incidence of Death
Description: Number of deaths within 90 days of the procedure.
Time Frame: with 90 days of the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
Number analyzed (Participants) | 61 | 68
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: within 24 hours of procedure
Arm/Group | Adenosine and Isoproterenol | Isoproterenol
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/68
Serious Adverse Events (participants affected / at risk) | 4/61 | 3/68
Other Adverse Events (participants affected / at risk) | 0/61 | 0/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Adenosine and Isoproterenol (N=61) | Isoproterenol (N=68)
Site hematoma (Vascular disorders) | 2 | 2 — Femoral vein/groin hematoma.
Pericardial Effusion (Vascular disorders) | 1 | 0 — Pericardial effusion with hemodynamic compromise.
A V Fistula (Vascular disorders) | 1 | 0 — Arterio venous fistula between femoral artery and vein.
Transient phrenic nerve paralysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 — Phrenic nerve paralysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes